CLINICAL TRIAL: NCT04887233
Title: Efficacy and Safety of Longan Extract Spray (P80 Spray) in Volunteers With Coronavirus Disease 2019 (COVID-19)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 214/64
Record Dates: First submitted 2021-05-13; First posted 2021-05-14 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Infection Viral
Keywords: Longan; nasal spray; COVID 19; efficacy; safety
MeSH Terms: conditions — Virus Diseases; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Longan nasal spray (Experimental): The patients will be received 2 puff of Longan nasal spray 2 times/day for 3 days.
  Interventions: Other: Longan nasal spray
- Placebo nasal spray (Placebo Comparator): The patients will be received 2 puff of placebo nasal spray 2 times/day for 3 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Longan nasal spray — The patients will be received 2 puff of Longan nasal spray 2 times/day for 3 days.
  Arms: Longan nasal spray
Other: Placebo — The patients will be received 2 puff of placebo nasal spray 2 times/day for 3 days.
  Arms: Placebo nasal spray

SUMMARY:
The objectives of this study are to evaluate efficacy and safety of longan extract spray (P80 spray) in volunteers with coronavirus disease 2019 (COVID19).Patients who infected COVID 19 (positive COVID 19 RT-PCR from nasal swab) are enrolled in the study. They will be treated with standard treatment of COVID 19. In addition, the patients will received longan extract nasal spray (P80 spray) or placebo nasal spray for 3 days (6 times). After that, they will be nasal swabbed for detecting COVID 19 infection. Adverse event will also be evaluated by physician or nurse.

DETAILED DESCRIPTION:
Patients who infected COVID 19 (positive COVID 19 RT-PCR from nasal swab) and pass inclusion criteria are enrolled in the study. The patients will be checked the clinical symptoms and chest x-ray by physician. They will be treated with standard treatment of COVID 19. In addition, the patients will received longan extract nasal spray (P80 spray) or placebo nasal spray for 3 days (6 times). Physician or nurse will ask for adverse events every day. After 3 days, the patients will be nasal swabbed for detecting COVID 19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Positive nasal swab test of coronavirus disease 2019 (COVID-19) (reverse transcriptase-polymerase chain reaction (RT-PCR) เป็นบวก (cycle threshold <40))
* Mild symptom with normal chest radiograph
* No history of Chronic Obstructive Pulmonary Disease (COPD) and other chronic lung diseases, Chronic kidney disease (CKD), Cardiovascular diseases and congenital heart diseases, Cerebrovascular diseases, Poorly controlled diabetes,BMI > 35 kg/m2, Cirrhosis, Immunocompromised condition
* Can read and write
* Vulnerable to participate

Exclusion Criteria:

* Allergic history to longan
* Uncontrollable disease status
* Pregnancy or lactation
* Participated in other studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Nasal swab test negative | 3 days
  There will be a negative reverse transcriptase-polymerase chain reaction (RT-PCR) test

SECONDARY OUTCOMES:
Absent of respiratory symptoms | 3 days
  There will be a body temperature less than 37.5 degree celsius and absent of respiratory symptoms.
No adverse event | 3 days
  There will be no allergic reaction

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Ph.D, Study Director — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: No